CLINICAL TRIAL: NCT07092176
Title: Randomized Controlled Study on Fall Prevention in Community-Dwelling Older Adults: Physiatry Based Steady Strides Intervention vs Primary Care
Brief Title: Steady Stride Fall Prevention Protocol vs Standard of Care
Acronym: SteadyStrides
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steady Strides: Fall Prevention and Stroke Rehabilitation Medical Institute (Industry)
Responsible Party: Principal Investigator, Levan Atanelov, CEO and Practice Owner, Steady Strides: Fall Prevention and Stroke Rehabilitation Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSRCT1
Record Dates: First submitted 2025-01-14; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Fall Prevention; Falls
Keywords: Falls; Fall Risk; Physiatry; Physical Therapy; Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Baseline assessment is masked, and outcomes assessment is if not fully, at least partially masked. Full masking can't be ensured for outcomes assessor and care providers as participants are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in the control arm will receive a one-time assessment by a trained research assistant at baseline and once more at 2 month follow up. Research assistant will measure and document the specified demographic and clinical variables to be compared between the control and intervention groups.
  The usual care will be provided as per the primary care provider's discretion. Providers will be advised to complete the CDC's STEADI (Stopping Elderly Accidents, Deaths, and Injuries) tool via CDC's training portal.
- Steady Strides (Experimental): Steady Strides Fall Prevention Protocol. See below for more detail.
  Interventions: Other: Steady Strides

INTERVENTIONS:
Other: Steady Strides — Participants in the control arm will receive a one-time assessment by a trained research assistant at baseline and once more at 2 month follow up. Research assistant will measure and document the specified demographic and clinical variables to be compared between the control and intervention groups.
  Participants in the intervention arm will receive a multifactorial intervention, including: Medical Intervention: Provided by physician(s) and/or nurse practitioners (NPs) or physician assistants (PAs) trained in the Steady Strides fall prevention protocol via the hybrid online and in person course on the Steady Strides fall prevention protocol . Rehabilitation Intervention: Provided by occupational therapists (OTs) and physical therapists (PTs) trained through a hybrid online and in person course on the Steady Strides fall prevention protocol
  Arms: Steady Strides

SUMMARY:
Falls are the leading cause of preventable morbidity and mortality in community dwelling older US adults (65 years old and older) . This is a research study to evaluate the comparative effectiveness of the structured physiatry-based Steady Strides Fall Prevention Protocol compared to the standard of care treatment provided by primary care providers in preventing falls in community-dwelling older adults.

DETAILED DESCRIPTION:
1. Background/Literature Review 1.1 Background Falls are the leading cause of preventable morbidity and mortality in community dwelling older US adults (65 years old and older) . This is a research study to evaluate the comparative effectiveness of the structured physiatry-based Steady Strides Fall Prevention Protocol compared to the standard of care treatment in preventing falls in community-dwelling older adults. Current standard of care is for the primary care physicians to evaluate patients at risk of falls, order medical work up, specialist physician consultation(s), medication changes and other interventions as needed, and prescribe physical and/or occupational therapy. Widely publicized guidelines for primary care physicians managing older adults at risk of falls include the American Geriatrics Society (3) and/or the Center for Disease Control and Prevention Stopping Elderly Accidents Deaths and Injuries (STEADI) guidelines. The American Geriatrics Society recommends that older adults undergo annual fall risk screening by physicians , which is an essential component of the annual Medicare wellness visit . To support a structured approach for physician-led fall prevention, the Centers for Disease Control and Prevention's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative provides an algorithmic framework for identifying, risk stratifying, and managing older adults at risk for falls, specifically designed for primary care providers . The STEADI algorithm includes evaluations of fall frequency, fear of falling, assessments for postural hypotension, foot deformities, visual and cognitive deficits, a basic screen for balance and gait issues, and a review of medications that could increase fall risk . Importantly, the STEADI approach positions physicians as key leaders in fall prevention management, utilizing physical therapy, community evidence-based fall prevention programs, podiatry and other referrals as part of a comprehensive, multifactorial intervention protocol . Limited non-randomized data suggest that implementing the STEADI strategy in primary care settings can reduce fall-related hospitalizations . The intervention arm of the Steady Strides Protocol includes both standard care and a structured fall prevention program. The Steady Strides Protocol is not an experimental treatment, it has been practiced at our clinic for several years already and has been paid for by the insurance providers as regular physiatry and rehabilitation care since 2017.Steady Strides Fall Prevention Protocol has been already shown in retrospective studies to have significant efficacy in preventing falls in community dwelling older adults . Novelty of the protocol lies not in introducing new rehabilitation techniques but in translating evidence-based interventions into a structured, consistent and easily adoptable framework for clinical practice. Since systematic reviews consistently highlight the efficacy of functional, multifactorial interventions-such as exercise, environmental modifications, and comprehensive assessments-in mitigating fall risk ; Steady Strides Protocol includes utilizing multidisciplinary interventions using physical and occupational therapy providers working closely with physiatry providers and emphasizes close communication between the rehabilitation professionals to ensure optimal patient outcomes. Since functional deficits like self-care and gait or balance impairments are common in those with high fall risk ; Steady Strides Protocol involves functional medicine professionals: physiatrists (also know as physical medicine and rehabilitation, or PM&R providers, mid-level and/or physician) to help evaluate and manage patient fall risk and barriers to rehabilitation, prescribe rehabilitation protocols and set rehabilitation-goals. Consistent with increased evidence that occupational therapy can help reduce falls ; Steady Strides protocol regularly promotes occupational therapy interventions. Since incorporating cognitive training together with physical therapy has been shown to reduce falls ; Steady Strides Protocol prescribes incorporating dual-tasking activities during rehabilitation. Since there is evidence that fear of falling is associated with increased fall risk ; Steady Strides Protocol systematically focuses on reducing fear of falling. To ensure consistency and reliability of care delivery Steady Strides Protocol uses a standardized hybrid on-line and in-person training for PM&R clinicians and rehabilitation therapy providers. This course educates on how to perform a structured falls related history, physical exam, interventions and a how to set standardized set of rehabilitation goals in order to identify and treat chronic biomechanical factors contributing to increased fall risk. Steady Strides Protocol also focuses on increased patient engagement consistent with general good clinical practice, as well as in context of emerging evidence that patient engagement may reduce fall risk .
2. Rationale/Significance/Problem Statement

   2.1 Rationale While the role of primary care providers in managing falls in older adults is crucial, investigators believe that fall prevention should primarily be managed by physicians trained in functional medicine, given that "medical reasons" are not the most common causes of falls. For example, one commonly thought of "medical reason" for falls, syncope, accounts for no more than 5% of falls in this population . Similarly, there is no strong association between falls and urinary tract infection, another commonly considered "medical reason" for falls in the elderly population. Whereas, by some estimates "mechanical falls," a term often used for "non-medical" causes, represent over 62% of falls among older adults presenting to emergency departments. Frequently reported causes of falls include slips, trips, and loss of balance, while factors often associated with falls include poor balance and difficulties with activities of daily living. Systematic reviews have consistently shown that functional, multifactorial interventions-such as exercise and environmental assessment and modification-are effective in preventing falls . It has been described that functional deficits, which serve as the final common pathway for various medical conditions, frequently constitute the majority of chronic predisposing risk factors for falls. These predisposing factors, such as gait and balance deficits, impaired vision, orthostatic hypotension, and impairments in cognitive function, Activity of Daily Living (ADLs), and Instrumental Activity of Daily Living (iADLs ), often play a significant role in increasing fall risk, with gait and balance problems frequently being the primary contributors. It therefore appears that functional deficits making up the final common pathway for different medical conditions often comprise the bulk of the chronic predisposing fall risk factors for falls . Given the strong evidence supporting functional medicine in fall prevention and the complexity of the neurological systems involved in balance and gait control , a biomechanical and functional assessment and treatment approach is preferred for managing older patients at risk of falls. Therefore, investigators advocate for a physiatrist-based approach for older adults at risk, as physiatrists specialize in functional medicine and the management of biomechanical impairments that affect human function, bridging functional and traditional medical approaches. Steady Strides is a structured, physiatrist-led, multifactorial functional assessment and management intervention. It combines a biomechanics-based functional physiatrist approach with comprehensive orthopedic, vestibular, podiatric, psychological, and neurological assessments to identify and treat the specific underlying biomechanical conditions that increase the risk of falls in older adults.

   2.2 Significance Steady Strides protocol efficacy was demonstrated in a retrospective chart review observational cohort study , but there are no previously published physiatry-based randomized controlled studies of structured fall prevention interventions. This is the first structured physiatry-based randomized controlled study for preventing falls in community dwelling older adults.
3. Study Purpose and Objectives 3.1 Purpose Aim: Falls are the leading cause of preventable morbidity and mortality in community dwelling older US adults (65 years old and older) . This is a research study to evaluate the comparative effectiveness of the structured physiatry-based Steady Strides Fall Prevention Protocol compared to the standard of care treatment in preventing falls in community-dwelling older adults. Current standard of care is for the primary care physicians to evaluate patients at risk of falls, order medical work up, specialist physician consultation(s), medication changes and other interventions as needed, and prescribe physical and/or occupational therapy. Widely publicized guidelines for primary care physicians managing older adults at risk of falls include the American Geriatrics Society and/or the Center for Disease Control and Prevention Stopping Elderly Accidents Deaths and Injuries (STEADI) guidelines. The intervention arm of the Steady Strides Protocol includes both standard care, that is follow up with the primary care and a structured physiatrist-led fall prevention program administered by licensed physical and occupational therapist providers with additional certification in utilizing the Steady Strides Fall Prevention Protocol. Physiatrist and therapist providers are trained using standardized hybrid in-person and online educational materials available at www.steadystridesacademy.com. This training is to standardize education and delivery of service of the Steady Strides Fall Prevention Protocol. Steady Strides Fall Prevention Protocol is not an experimental treatment and preliminary evidence from observational study with the protocol has shown good clinical outcomes.

3.2 Hypothesis: investigators hypothesize that participation in Steady Strides Fall Prevention Program will significantly reduce the number of falls compared to management by primary care providers as per standard of care.

3.3 Objectives

Primary Objective:

To evaluate the effectiveness of the Steady Strides protocol in reducing falls among community dwelling older adults six months after the intervention, specifically targeting individuals who have reported at least two falls in the previous six months.

Secondary Objectives: To evaluate the impact of the intervention on fall-related morbidity and mortality, the rate of hospitalizations, emergency department (ED) visits and other health-care utilization. To assess the impact of the intervention on reduction in fall rates from baseline; fall risk, ADLs, frailty, fear of falls, community integration, cognitive function, sleep and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants must be community-dwelling older adults aged 65 years or older.

Fall History: Participants must have reported experiencing at least two falls in the six months prior to the intake visit.

Independence: Participants must report the ability to drive independently at the time of the intake visit and ambulate at least 10 feet with or without an assistive device (e.g. cane or walker, wheelchair ambulators are not included). Participants must report their ability to independently make medical decisions and sign their medical paperwork, including consent to participate in the study.

Setting: Participants must reside in a community setting, not in a long-term care facility or hospital.

Language: Participants must report ability to speak, read and comprehend English fluently.

Exclusion Criteria: No additional exclusion criteria beyond those specified in the inclusion criteria. All individuals who meet the inclusion criteria are eligible to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Falls | Total falls reported after completion of the intervention 6 months after the intervention.
  The primary outcome is self-reported total number of falls during the 6 months of the follow up period after the 2 month intervention. Values 0-100. Lower number are better functioning.
  Falls were defined as "unintentionally coming to the ground or some lower level and other than as a consequence of sustaining a violent blow, loss of consciousness, sudden onset of paralysis as in stroke or an epileptic seizure."

SECONDARY OUTCOMES:
Fall-Related Morbidity-number of hospitalizations or ED visits | assessed monthly at months 1-8
  number of hospitalizations or ED visits. Possible values 0-100, lower number better function.
Fall Risk | Assessed at the completion of the intervention (2 months after the first visit)
  Assessed using Single Leg Stance. Seconds, 0-100. Higher numbers are better
Fall-Related Healthcare Utilization | baseline and monthly for 8 months
  Self reported number of Days in Hospital or in Nursing Home/Subacute Rehab Facility due to falls in the past month.
  values 0-100, less is better functioning.
Fear of Falls | Assessed at the completion of the intervention (2 months after the first visit)
  FES-I (Falls Efficacy Scale - International): Measures fear of falling during daily activities. Values 16-64, lower numbers are better functioning
iADLs | Assessed at the completion of the intervention (2 months after the first visit)
  Lawton Instrumental Activities of Daily Living Scale: Assesses ability to perform daily tasks such as shopping, managing finances, and preparing meals. Scale 0-8, higher number better functioning.
Functional Reach Test | at baseline and at month 2
  Functional Reach Test assesses fall risk in context of functional reach, e.g. during ADLs. 0-20 inches. higher number is better functioning.
Frailty | Assessed at the completion of the intervention (2 months after the first visit)
  Clinical Frailty Scale used to assess. 1-9, lower number is better functioning.
General cognitive function | Assessed at the completion of the intervention (2 months after the first visit)
  MOCA (Montreal Cognitive Assessment): Screens for mild cognitive impairment. Scores 0-30, higher number is better functioning.
Cognitive Flexibility | Assessed at the completion of the intervention (2 months after the first visit)
  Trail Making Test (Parts A and B): Assesses cognitive flexibility and set-shifting ability. 0-300 seconds, lower number is better functioning.
Anxiety | Assessed at the completion of the intervention (2 months after the first visit)
  GAD-7 (Generalized Anxiety Disorder Scale): Screens for generalized anxiety symptoms. Scores 0-21, lower number is better functioning.
Depression | Assessed at the completion of the intervention (2 months after the first visit)
  GDS-15 (Geriatric Depression Scale): Screens for depressive symptoms. Score 0-15, lower function is better functioning.
Sleepiness | Assessed at baseline and month 2
  Epworth Sleepiness Scale Short Form 8. Score 0-24, lower number is better functioning.
Home Safety as a risk factor for falls | At baseline and 2 months
  Home Safety Assessment Tool. Standardized tool, scores 0-74, lower number is a safer home for fall risk
Community Integration | Baseline and 2 months follow up
  Community Integration Questionnaire - Revised (CIQ-R). score 0-29, lower number is better functioning.
Fall related morbidity-fall severity | 0-8 months
  Mild: Number of falls causing no pain or pain lasting < 1 hour in the past month-values 0-100 Moderate: Number of falls causing pain lasting for at least 1 hour and/or causing bruising in the past month-values 0-100 Severe: Number of falls causing fractures or head trauma in the past month-values 0-100 Lower number is better functioning.
Fall Risk-TUG | baseline and 2 months
  Timed Up and Go Test , lower number are better, 0-100 sec .
Side Effects Severity | baseline through month 8
  Count 0-100 of number of adverse events associated with rehabilitation. Lower number is better Mild: Number Events Causing Pain or Bruising lasting < 1 hour , occurred while doing Rehab in the past month Moderate: Number of Events Causing Pain or Bruising lasting more than 1 hour , occurred while doing Rehab in the past month Severe: Number of Events Causing Head Trauma , occurred while doing Rehab in the past month Severe: number of Events Causing Fracture(s) , occurred while doing Rehab in the past month

CONTACTS AND LOCATIONS:
Locations (1):
- Steady Strides, Owings Mills, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ha VT, Nguyen TN, Nguyen TX, Nguyen HTT, Nguyen TTH, Nguyen AT, Pham T, Vu HTT. Prevalence and Factors Associated with Falls among Older Outpatients. Int J Environ Res Public Health. 2021 Apr 12;18(8):4041. doi: 10.3390/ijerph18084041. PMID 33921355
- [Background] Kakara R, Bergen G, Burns E, Stevens M. Nonfatal and Fatal Falls Among Adults Aged >/=65 Years - United States, 2020-2021. MMWR Morb Mortal Wkly Rep. 2023 Sep 1;72(35):938-943. doi: 10.15585/mmwr.mm7235a1. PMID 37651272
- [Background] Guideline for the prevention of falls in older persons. American Geriatrics Society, British Geriatrics Society, and American Academy of Orthopaedic Surgeons Panel on Falls Prevention. J Am Geriatr Soc. 2001 May;49(5):664-72. No abstract available. PMID 11380764
- [Background] The prevention of falls in later life. A report of the Kellogg International Work Group on the Prevention of Falls by the Elderly. Dan Med Bull. 1987 Apr;34 Suppl 4:1-24. PMID 3595217
- [Background] Phelan EA, Mahoney JE, Voit JC, Stevens JA. Assessment and management of fall risk in primary care settings. Med Clin North Am. 2015 Mar;99(2):281-93. doi: 10.1016/j.mcna.2014.11.004. PMID 25700584
- [Background] Stevens JA, Smith ML, Parker EM, Jiang L, Floyd FD. Implementing a Clinically Based Fall Prevention Program. Am J Lifestyle Med. 2017 Jul 5;14(1):71-77. doi: 10.1177/1559827617716085. eCollection 2020 Jan-Feb. PMID 31903086
- [Background] Johnston YA, Bergen G, Bauer M, Parker EM, Wentworth L, McFadden M, Reome C, Garnett M. Implementation of the Stopping Elderly Accidents, Deaths, and Injuries Initiative in Primary Care: An Outcome Evaluation. Gerontologist. 2019 Nov 16;59(6):1182-1191. doi: 10.1093/geront/gny101. PMID 30239774
- [Background] Tricco AC, Thomas SM, Veroniki AA, Hamid JS, Cogo E, Strifler L, Khan PA, Robson R, Sibley KM, MacDonald H, Riva JJ, Thavorn K, Wilson C, Holroyd-Leduc J, Kerr GD, Feldman F, Majumdar SR, Jaglal SB, Hui W, Straus SE. Comparisons of Interventions for Preventing Falls in Older Adults: A Systematic Review and Meta-analysis. JAMA. 2017 Nov 7;318(17):1687-1699. doi: 10.1001/jama.2017.15006. PMID 29114830
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Guirguis-Blake JM, Michael YL, Perdue LA, Coppola EL, Beil TL. Interventions to Prevent Falls in Older Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Apr 24;319(16):1705-1716. doi: 10.1001/jama.2017.21962. PMID 29710140
- [Background] Ganz DA, Latham NK. Prevention of Falls in Community-Dwelling Older Adults. N Engl J Med. 2020 Feb 20;382(8):734-743. doi: 10.1056/NEJMcp1903252. No abstract available. PMID 32074420
- [Background] Chu MM, Fong KN, Lit AC, Rainer TH, Cheng SW, Au FL, Fung HK, Wong CM, Tong HK. An Occupational Therapy Fall Reduction Home Visit Program for Community-Dwelling Older Adults in Hong Kong After an Emergency Department Visit for a Fall. J Am Geriatr Soc. 2017 Feb;65(2):364-372. doi: 10.1111/jgs.14527. Epub 2016 Nov 17. PMID 27858951
- [Background] Liu M, Xue QL, Gitlin LN, Wolff JL, Guralnik J, Leff B, Szanton SL. Disability Prevention Program Improves Life-Space and Falls Efficacy: A Randomized Controlled Trial. J Am Geriatr Soc. 2021 Jan;69(1):85-90. doi: 10.1111/jgs.16808. Epub 2020 Sep 20. PMID 32951215
- [Background] Nascimento MM, Maduro PA, Rios PMB, Nascimento LDS, Silva CN, Kliegel M, Ihle A. The Effects of 12-Week Dual-Task Physical-Cognitive Training on Gait, Balance, Lower Extremity Muscle Strength, and Cognition in Older Adult Women: A Randomized Study. Int J Environ Res Public Health. 2023 Apr 13;20(8):5498. doi: 10.3390/ijerph20085498. PMID 37107780
- [Background] Pang MYC, Yang L, Ouyang H, Lam FMH, Huang M, Jehu DA. Dual-Task Exercise Reduces Cognitive-Motor Interference in Walking and Falls After Stroke. Stroke. 2018 Dec;49(12):2990-2998. doi: 10.1161/STROKEAHA.118.022157. PMID 30571419
- [Background] Strouwen C, Molenaar EALM, Munks L, Keus SHJ, Zijlmans JCM, Vandenberghe W, Bloem BR, Nieuwboer A. Training dual tasks together or apart in Parkinson's disease: Results from the DUALITY trial. Mov Disord. 2017 Aug;32(8):1201-1210. doi: 10.1002/mds.27014. Epub 2017 Apr 25. PMID 28440888
- [Background] Gambaro E, Gramaglia C, Azzolina D, Campani D, Molin AD, Zeppegno P. The complex associations between late life depression, fear of falling and risk of falls. A systematic review and meta-analysis. Ageing Res Rev. 2022 Jan;73:101532. doi: 10.1016/j.arr.2021.101532. Epub 2021 Nov 27. PMID 34844015
- [Background] Asai T, Oshima K, Fukumoto Y, Yonezawa Y, Matsuo A, Misu S. The association between fear of falling and occurrence of falls: a one-year cohort study. BMC Geriatr. 2022 May 5;22(1):393. doi: 10.1186/s12877-022-03018-2. PMID 35509040
- [Background] Dykes PC, Carroll DL, Hurley A, Lipsitz S, Benoit A, Chang F, Meltzer S, Tsurikova R, Zuyov L, Middleton B. Fall prevention in acute care hospitals: a randomized trial. JAMA. 2010 Nov 3;304(17):1912-8. doi: 10.1001/jama.2010.1567. PMID 21045097
- [Background] Rubenstein LZ, Josephson KR. The epidemiology of falls and syncope. Clin Geriatr Med. 2002 May;18(2):141-58. doi: 10.1016/s0749-0690(02)00002-2. PMID 12180240
- [Background] Rowe T, Towle V, Van Ness PH, Juthani-Mehta M. Lack of positive association between falls and bacteriuria plus pyuria in older nursing home residents. J Am Geriatr Soc. 2013 Apr;61(4):653-4. doi: 10.1111/jgs.12177. No abstract available. PMID 23581923
- [Background] Sri-on J, Tirrell GP, Lipsitz LA, Liu SW. Is there such a thing as a mechanical fall? Am J Emerg Med. 2016 Mar;34(3):582-5. doi: 10.1016/j.ajem.2015.12.009. Epub 2015 Dec 12. PMID 26795891
- [Background] Lord SR, Ward JA, Williams P, Anstey KJ. An epidemiological study of falls in older community-dwelling women: the Randwick falls and fractures study. Aust J Public Health. 1993 Sep;17(3):240-5. doi: 10.1111/j.1753-6405.1993.tb00143.x. PMID 8286498
- [Background] Horak FB. Postural orientation and equilibrium: what do we need to know about neural control of balance to prevent falls? Age Ageing. 2006 Sep;35 Suppl 2:ii7-ii11. doi: 10.1093/ageing/afl077. PMID 16926210
- See also: Centers for Disease Control and Prevention. STEADI: Provider Training & Continuing Education — https://www.cdc.gov/steadi/hcp/training/index.html
- See also: Aaron David Abrishami, Aviel Hanasab, Eliot Sadik, et al. Efficacy of Steady Strides: A Structured Physiatrist-Led Intervention for Reducing Falls in High-Risk Ambulatory Community Dwelling Older Adults: An Observational Cohort Study. . J Med - Clin Res — https://www.scivisionpub.com/pdfs/efficacy-of-steady-strides-a-structured-physiatristled-intervention-for-reducing-falls-in-highrisk-ambulatory-communitydwelling-ol-3062.pdf
- See also: Centers for Medicare & Medicaid Services (CMS). Medicare wellness visits — https://www.cms.gov/Outreach-and-Education/Medicare-Learning-Network-MLN/MLNProducts/preventive-services/medicare-wellness-visits.html
- See also: Centers for Disease Control and Prevention. Algorithm for Fall Risk Screening, Assessment, and Intervention. Centers for Disease Control and Prevention 2012 — https://www.cdc.gov/steadi/media/pdfs/STEADI-Algorithm-508.pdf
- See also: Atanelov L. Steady Strides Fall Prevention Training Course. 2025 — https://steadystridesacademy.com/course/steady-strides-fall-prevention-training-course